CLINICAL TRIAL: NCT04532671
Title: Evaluation of Clinical Performance of 3D Printed Polyether Ether Ketone (PEEK) Inlays Compared With Milled Indirect PEEK Inlays Versus Indirect Resin Composite Inlays Over One Year Period of Time (A Randomized Clinical Trial)
Brief Title: Evaluation of Clinical Performance of 3D Printed Polyether Ether Ketone (PEEK) Inlays
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, donia elshafey, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 88245
Record Dates: First submitted 2020-08-17; First posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Occlusal Caries
MeSH Terms: interventions — poly(phthalazine ether sulfone ketone)

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Poly ether ether ketone (PEEK) (Other): Poly ether ether keton (PEEK) is acknowledged as a high-performance polymer in engineering & medical applications due to its favorable mechanical and chemical properties.
  Interventions: Other: Poly ether ether ketone (PEEK)
- CADCAM poly ether ether ketone (PEEK) (Other): PEEK was predominantly processed out of CAD/CAM-supported milled out of prefabricated blanks.
  Interventions: Other: CADCAM Poly ether ether ketone (PEEK)
- indirect resin composite (Active Comparator): In CAD/CAM resin composite blocks, properties of flexibility and ease of use similar to that of resin composite are combined with durability and surface finish properties similar to that of ceramics
  Interventions: Other: indirect resin composite

INTERVENTIONS:
Other: Poly ether ether ketone (PEEK) — PEEK has been used in dentistry so far in certain fields as for, removable and fixed dental prostheses, implants, and implant abutments as well as orthodontic devices, whereas in literature, it is mostly mentioned in relation to prosthetics. PEEK was predominantly processed out of CAD/CAM-supported milled out of prefabricated blanks. Producing dental restorations via Additive manufacturing is still hardly widespread
  Arms: Poly ether ether ketone (PEEK)
Other: CADCAM Poly ether ether ketone (PEEK) — Increased demand for long-lasting restoration's properties have led to many improvements in the production techniques of posterior restorations such as CAD/CAM systems. This technique simplifies the production of indirect restorations and make it possible to use advanced materials as PEEK
  Arms: CADCAM poly ether ether ketone (PEEK)
Other: indirect resin composite — CADCAM resin composite blocks using milling process
  Arms: indirect resin composite

SUMMARY:
In patients using Inlay restorations will the use of 3D printed PEEK material and technique have superior clinical performance to milled PEEK one or to milled composite resin inlays, evaluation of restorations will be done at baseline, six months and 12 months using the modified US Public Health Service (USPHS) evaluation system

DETAILED DESCRIPTION:
The study will be conducted in Conservative Dentistry Department, Faculty of Dentistry, Cairo University; The operator in charge will be Donia Mamdouh Elshafey Patients will be selected from the outpatient clinic of the department Conservative Dentistry Department, Faculty of Dentistry, Cairo University All cavity preparations will be performed with fine inlay burs according to inlay cavity principles. The walls facing each other will be prepared 5 to 6 degree divergent with 80 μm diamond burs and were finished with 25 μm diamond burs. All internal angles will be rounded and all edges will terminate in the enamel. The pulpal floor will be prepared at a depth of at least 1.5 mm. The teeth will be discarded if isthmus width was more than 2/3 of the distance between the tubercule tips, or if the walls are thinner than 2 mm before the preparation or thinner than 1.5 mm after the preparation. The caries affected dentin tissue at the cavity floor will be left. The teeth will be discarded from study if the pulp is exposed. To eliminate irregular areas in the cavities, a liner will be applied as a blockout material. Then the operator will adhere strictly to the manufacturer's instructions in the imaging, computer design and machining of the restorations either 3D printing or milling procedure.

The prepared teeth for the indirect restorations will be scanned with an optical 3D camera (CEREC Omnicam, Dentsply Sirona, Bensheim, Germany), inlays will be designed by a CAD software (CEREC SW 4.6.1, Dentsply Sirona), and files will be created in STL format (inLab CAD SW 18.1, Dentsply Sirona) then inlays will additively manufactured After the printing process is finished, the inlays will be immediately removed from the building platform and cooled down at room temperature. The inlay will be adapted individually to its cavity, and the occlusal surface will be recontoured. Such post processing also will be performed on the milled inlays. After all inlays are adequately adapted, they will be adhesively inserted into the cavities.

ELIGIBILITY:
Inclusion Criteria:

* Patients aging greater than or equal 18 years.
* Patients with a high level of oral hygiene.
* Each patient enrolled in the study had moderate to large size carious lesion or defective restoration to be replaced on a maxillary or mandibular permanent molar.
* Patients with good likelihood of recall availability.

Exclusion Criteria:

* Participants with general/systemic illness.
* Pregnant or lactating females.
* Concomitant participation in another research study.
* Inability to comply with study procedures.
* Heavy bruxism habits.
* Last experience with allergic reactions against any components of the used materials.
* Patients receiving orthodontic treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Marginal integrity | 12 months
  Visual inspection with explorer and mirror, Distance penetrated by the Explorer at the tooth restoration interface
marginal discoloration | 12 months
  Visual inspection with a mirror at 18 inches, the degree of mismatch from the normal range of tooth shades and translucency Visual inspection to check the proximity of the shade from the natural tooth
secondary caries | 12 months
  Visual inspection of discoloration that occurs on the tooth after the filling has been used for a period of time
post operative sensitivity | 12 months
  Asking the patient if there is any associated pain after adding the restoration

CONTACTS AND LOCATIONS:
Overall Officials: Donia M elshafey, master, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: Yes
Undecided: It is not yet known if there will be a plan to make IPD available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: expecting to have all the data during october 2022
Access Criteria: IPD through contacting the main author doniamamdouh@dentistry.cu.edu.eg.com
URL: http://erepository.cu.edu.eg/index.php/cutheses